CLINICAL TRIAL: NCT02248142
Title: Sifrol® (Pramipexole) Impact on RLS: A 12-weeks Observational Study in Patients With Primary RLS
Brief Title: Observational Study of Sifrol® in Patients With Primary Restless Legs Syndrome (RLS)
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 248.623
Record Dates: First submitted 2014-09-22; First posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Pramipexole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- RLS patients
  Interventions: Drug: Pramipexole

INTERVENTIONS:
Drug: Pramipexole
  Other Names: Sifrol®

SUMMARY:
Study to evaluate treatment effect of pramipexole on RLS severity as measured by IRLS, CGI-I and RLS-6 and to evaluate the time needed to reach maintenance dose of Pramipexole (PPX)

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from primary RLS who are planned to be initiated on treatment with pramipexole as part of the routine care could be included into the study
* Patients not pre-treated with any dopaminergic agent (de novo patients) or patients pretreated with dopaminergic medication
* Male or female patients of any age

Exclusion Criteria:

* Treating physicians are asked to consider the regulations described in the Summary of Product Characteristics (SPC) for the treatment with pramipexole

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients suffering from moderate to severe RLS recruited at office-based neurologists
Sampling Method: Non-Probability Sample
Enrollment: 1029 (Actual)
Dates: Start 2006-02; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Assessment of RLS symptoms (IRLS) on a 4-point rating scale | up to 12 weeks
Assessment of RLS severity on a 6-point rating scale | up to 12 weeks

SECONDARY OUTCOMES:
Change in Clinical Global Impression Improvement (CGI-I) rated on a 7-point scale | up to 12 weeks
Global assessment of efficacy by investigator on a 5-point scale | after 12 weeks
Number of patients with adverse events | up to 12 weeks
Time to reach maintenance dose of pramipexole | up to 12 weeks